CLINICAL TRIAL: NCT01405430
Title: Exploration of New Biologic Factors' Predictive Value , Especially Circulating VE-cadherin in Metastatic Colorectal Adenocarcinoma Patients Treated With Bevacizumab
Brief Title: Exploration of Circulating VE-cadherin in Metastatic Colorectal Adenocarcinoma Patients Treated With Bevacizumab
Acronym: AVECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: UMR-S Inserm 1036 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AVECC; ET2010-003 (Other: Sponsor's identification)
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer; Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + blood samples (Experimental)
  Interventions: Biological: Bevacizumab + blood samples

INTERVENTIONS:
Biological: Bevacizumab + blood samples — Bevacizumab will be administered according to investigators appreciation.
  Blood samples will be collected at enrollment, at second bevacizumab's administration and every 10 weeks until progression, or until patients stop bevacizumab because of toxicity or until one year at most in case that patients still receive bevacizumab.

SUMMARY:
It is a prospective, non-randomized, monocentric study. The purpose of the study is to assess the predictive value of VE-cadherin on the objective tumor response.

Biological factors will be correlated to clinical outcome measures.

100 patients treated with bevacizumab for a metastatic colorectal adenocarcinoma will be enrolled.

Patients will be followed every 10 weeks until progression in spite of bevacizumab or until they stop bevacizumab because of toxicity.

Bevacizumab will be administered according to investigators appreciation.

Blood samples will be collected at enrollment, at second bevacizumab's administration and every 10 weeks until progression, or until patients stop bevacizumab because of toxicity or until one year at most in case that patients still receive bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a metastatic colorectal cancer proved histologically and treated with bevacizumab in first line.
* At least one extra-osseous, non-irradiated, measurable site (>= 10 mm with spiral CT).
* No prior radiotherapy treatment unless treatment is over for at least 4 weeks.
* Adult patients.
* PS <= 2.
* Life expectancy greater than 3 months.
* Mandatory affiliation with a healthy security insurance.
* Signed written informed consent.

Exclusion Criteria:

* Prior chemotherapy for the metastatic cancer.
* Prior bevacizumab treatment.
* Other current cancer or previous cancer detected in the last 5 years that can be linked to the current disease.
* Patient deprived of freedom.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Response rate to treatment | Up to 1 year at most
  A 30% response rate (complete or partial response) to treatment is expected. The response will be assessed according to RECIST criteria. This primary outcome measure is defined by the observation of at least one objective response during the treatment.
  This outcome measure will be correlated to biological factors.

SECONDARY OUTCOMES:
Clinical benefit | At progression or up to 1 year at most
  The clinical benefit is based on complete response, partial response or stable disease.
  This outcome measure will be correlated to biological factors.
Evaluation of progression-free survival | From the beginning of treatment to progression, death or last available information
  This outcome measure will be correlated to biological factors.
Evaluation of overall survival | From the beginning of treatment to death or last available information
  This outcome measure will be correlated to biological factors.
Evaluation of tumoral markers | At progression with bevacizumab or up to 1 year of follow-up at most
  Evaluation of ACE and Ca19-9
Evaluation of vascular toxicities | Up to 1 year
  Assess the link between vascular toxicities and VE-cadherin rate. These toxicities will be assessed during the follow-up of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle DE LA FOUCHARDIERE, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Hôpital Privé Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon

REFERENCES:
- [Background] Bouvier AM, Remontet L, Jougla E, Launoy G, Grosclaude P, Buemi A, Tretarre B, Velten M, Dancourt V, Menegoz F, Guizard AV, Mace Lesec'h J, Peng J, Bercelli P, Arveux P, Esteve J, Faivre J. Incidence of gastrointestinal cancers in France. Gastroenterol Clin Biol. 2004 Oct;28(10 Pt 1):877-81. doi: 10.1016/s0399-8320(04)95152-4. PMID 15523225
- [Background] Weitz J, Koch M, Debus J, Hohler T, Galle PR, Buchler MW. Colorectal cancer. Lancet. 2005 Jan 8-14;365(9454):153-65. doi: 10.1016/S0140-6736(05)17706-X. PMID 15639298
- [Background] Kozloff M, Yood MU, Berlin J, Flynn PJ, Kabbinavar FF, Purdie DM, Ashby MA, Dong W, Sugrue MM, Grothey A; Investigators of the BRiTE study. Clinical outcomes associated with bevacizumab-containing treatment of metastatic colorectal cancer: the BRiTE observational cohort study. Oncologist. 2009 Sep;14(9):862-70. doi: 10.1634/theoncologist.2009-0071. Epub 2009 Sep 2. PMID 19726453
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Background] Gruenberger B, Tamandl D, Schueller J, Scheithauer W, Zielinski C, Herbst F, Gruenberger T. Bevacizumab, capecitabine, and oxaliplatin as neoadjuvant therapy for patients with potentially curable metastatic colorectal cancer. J Clin Oncol. 2008 Apr 10;26(11):1830-5. doi: 10.1200/JCO.2007.13.7679. PMID 18398148
- [Background] Kabbinavar FF, Hambleton J, Mass RD, Hurwitz HI, Bergsland E, Sarkar S. Combined analysis of efficacy: the addition of bevacizumab to fluorouracil/leucovorin improves survival for patients with metastatic colorectal cancer. J Clin Oncol. 2005 Jun 1;23(16):3706-12. doi: 10.1200/JCO.2005.00.232. Epub 2005 May 2. PMID 15867200
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Kabbinavar FF, Schulz J, McCleod M, Patel T, Hamm JT, Hecht JR, Mass R, Perrou B, Nelson B, Novotny WF. Addition of bevacizumab to bolus fluorouracil and leucovorin in first-line metastatic colorectal cancer: results of a randomized phase II trial. J Clin Oncol. 2005 Jun 1;23(16):3697-705. doi: 10.1200/JCO.2005.05.112. Epub 2005 Feb 28. PMID 15738537
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Jain RK, Duda DG, Willett CG, Sahani DV, Zhu AX, Loeffler JS, Batchelor TT, Sorensen AG. Biomarkers of response and resistance to antiangiogenic therapy. Nat Rev Clin Oncol. 2009 Jun;6(6):327-38. doi: 10.1038/nrclinonc.2009.63. PMID 19483739
- [Background] Jubb AM, Hurwitz HI, Bai W, Holmgren EB, Tobin P, Guerrero AS, Kabbinavar F, Holden SN, Novotny WF, Frantz GD, Hillan KJ, Koeppen H. Impact of vascular endothelial growth factor-A expression, thrombospondin-2 expression, and microvessel density on the treatment effect of bevacizumab in metastatic colorectal cancer. J Clin Oncol. 2006 Jan 10;24(2):217-27. doi: 10.1200/JCO.2005.01.5388. Epub 2005 Dec 19. PMID 16365183
- [Background] Burstein HJ, Chen YH, Parker LM, Savoie J, Younger J, Kuter I, Ryan PD, Garber JE, Chen H, Campos SM, Shulman LN, Harris LN, Gelman R, Winer EP. VEGF as a marker for outcome among advanced breast cancer patients receiving anti-VEGF therapy with bevacizumab and vinorelbine chemotherapy. Clin Cancer Res. 2008 Dec 1;14(23):7871-7. doi: 10.1158/1078-0432.CCR-08-0593. PMID 19047116
- [Background] Schneider BP, Wang M, Radovich M, Sledge GW, Badve S, Thor A, Flockhart DA, Hancock B, Davidson N, Gralow J, Dickler M, Perez EA, Cobleigh M, Shenkier T, Edgerton S, Miller KD; ECOG 2100. Association of vascular endothelial growth factor and vascular endothelial growth factor receptor-2 genetic polymorphisms with outcome in a trial of paclitaxel compared with paclitaxel plus bevacizumab in advanced breast cancer: ECOG 2100. J Clin Oncol. 2008 Oct 1;26(28):4672-8. doi: 10.1200/JCO.2008.16.1612. PMID 18824714
- [Background] Willett CG, Boucher Y, di Tomaso E, Duda DG, Munn LL, Tong RT, Chung DC, Sahani DV, Kalva SP, Kozin SV, Mino M, Cohen KS, Scadden DT, Hartford AC, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Chen HX, Shellito PC, Lauwers GY, Jain RK. Direct evidence that the VEGF-specific antibody bevacizumab has antivascular effects in human rectal cancer. Nat Med. 2004 Feb;10(2):145-7. doi: 10.1038/nm988. Epub 2004 Jan 25. PMID 14745444
- [Background] Corada M, Zanetta L, Orsenigo F, Breviario F, Lampugnani MG, Bernasconi S, Liao F, Hicklin DJ, Bohlen P, Dejana E. A monoclonal antibody to vascular endothelial-cadherin inhibits tumor angiogenesis without side effects on endothelial permeability. Blood. 2002 Aug 1;100(3):905-11. doi: 10.1182/blood.v100.3.905. PMID 12130501
- [Background] Gory-Faure S, Prandini MH, Pointu H, Roullot V, Pignot-Paintrand I, Vernet M, Huber P. Role of vascular endothelial-cadherin in vascular morphogenesis. Development. 1999 May;126(10):2093-102. doi: 10.1242/dev.126.10.2093. PMID 10207135
- [Background] Wallez Y, Vilgrain I, Huber P. Angiogenesis: the VE-cadherin switch. Trends Cardiovasc Med. 2006 Feb;16(2):55-9. doi: 10.1016/j.tcm.2005.11.008. PMID 16473763
- [Background] Wallez Y, Cand F, Cruzalegui F, Wernstedt C, Souchelnytskyi S, Vilgrain I, Huber P. Src kinase phosphorylates vascular endothelial-cadherin in response to vascular endothelial growth factor: identification of tyrosine 685 as the unique target site. Oncogene. 2007 Feb 15;26(7):1067-77. doi: 10.1038/sj.onc.1209855. Epub 2006 Aug 14. PMID 16909109